CLINICAL TRIAL: NCT05322772
Title: A Study of Cardiac Arrhythmia and ECG Changes in Children With Convulsions at Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Eman Aiman Sadek, resident doctor at pediateric department sohag general hospital, Sohag University
Other Study IDs: Soh-Med-22-03-05
Record Dates: First submitted 2022-03-28; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Convulsions
MeSH Terms: conditions — Seizures | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- children with epilepsy: epilepsy diagnosed clinically EEG
  Interventions: Device: ECG
- children with febrile convulsions: the child has high grade fever from 6 month to 6 years not recurrent duration less than 15 minute or atypical febrile convulsions
  Interventions: Device: ECG
- children with cns infection: the child has fever, neck, rigidity DCL
  +or- CSF analysis
  Interventions: Device: ECG
- children with electrolyte imbalance, hypoglycemia: abnormal values of electrolyte hypoglycemia
  Interventions: Device: ECG
- children with poisoning: history of ingestion or inhalation of toxic substance
  Interventions: Device: ECG
- children with encephalopathy: the child complains of brain disease or mal function with altered mental status as a complication of primary illness as kidney failure ,cirrhosis, etc.
  Interventions: Device: ECG
- children with trauma: history of trauma imaging study done
  Interventions: Device: ECG
- children with genetic cause: the child has congenital anomaly as chromosomal abnormality, metabolic disease, mitochondrial disease
  Interventions: Device: ECG
- others: children not fulfilling the previous groups
  Interventions: Device: ECG

INTERVENTIONS:
Device: ECG — ii. 12 leads ECG: 12 leads ECG will be done to all infants & children using (FUKUDA DENSHI, CARDIMAX, model FCP 7101). The electrocardiograms will be reviewed through the creation of descriptive reports and determination of the following variables: heart rate, QRS duration, The QT interval was measured from the onset of the QRS complex to the end of the T wave, defined by the return of the terminal T wave to the isoelectric T-P baseline. When U waves were present, the end of the T wave will be taken as the nadir between the T and U waves. Then QT interval will be corrected for heart rate using Bazett's formula Interpretation of every ECG paper

SUMMARY:
Convulsion is a common pediatric disorder and there is strong relation between convulsion and cardiovascular system which revealed by ECG monitoring and there are many ECG abnormalities attributed to different causes of convulsions, A 12-lead ECG is a low-cost test and can detect clinically significant abnormalities such as long QTc interval or heart block. Doing an ECG in all patients presenting with seizures clinic, inevitably, pick up non-specific abnormalities which require further investigation. Moreover, a normal 12-lead ECG does not exclude a cardiovascular cause for collapse and for those in whom a cardiac cause is still suspected despite a normal ECG, referral to a cardiologist is advisable

ELIGIBILITY:
Inclusion Criteria:

* All children aged from 1month to 18 years presenting to the Pediatric Emergency with convulsions will be included.

Exclusion Criteria:

* Children not filling the criteria of convulsions (like conditions mimic epilepsy)
* Children with known cardiac disease or cardiac arrhythmia and patients who will not give consent will be excluded.

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All children aged from 1month to 18 years presenting to the Pediatric Emergency with convulsions will be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
heart rate | one year
  normal values according to age and sex.

SECONDARY OUTCOMES:
PR interval | one year
  normal values according to age and sex.

OTHER OUTCOMES:
QTC | one year
  normal values according to age and sex.

REFERENCES:
- [Background] Huang X, Malek N, Simpson J, Kalladka D, Dunn FG, Leach JP. Winning hearts and minds: ECG reporting in the first seizure clinic. BMC Cardiovasc Disord. 2021 Jul 31;21(1):364. doi: 10.1186/s12872-021-02174-4. PMID 34332536
- [Background] Rijnbeek PR, Witsenburg M, Szatmari A, Hess J, Kors JA. PEDMEANS: a computer program for the interpretation of pediatric electrocardiograms. J Electrocardiol. 2001;34 Suppl:85-91. doi: 10.1054/jelc.2001.28835. PMID 11781941
- [Background] Karjalainen J, Viitasalo M. Fever and cardiac rhythm. Arch Intern Med. 1986 Jun;146(6):1169-71. PMID 2424378